CLINICAL TRIAL: NCT00717548
Title: The Effectiveness of Narrative Exposure Therapy in Treating Women After Trafficking and Forced Prostitution
Brief Title: Efficacy of Narrative Exposure Therapy (NET) in Treating Women After Human Trafficking or Forced Prostitution
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Konstanz (Other)
Responsible Party: Principal Investigator, Martina Ruf, PhD, University of Konstanz
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FH05.06.2008
Record Dates: First submitted 2008-07-15; First posted 2008-07-17 (Estimated); Last update posted 2012-11-05 (Estimated); Status verified 2012-11

CONDITIONS: Posttraumatic Stress Disorder; Depression; Dissociation
Keywords: Somatic Complaints
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Dissociative Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Behavioral: Narrative Exposure Therapy

INTERVENTIONS:
Behavioral: Narrative Exposure Therapy — Trauma-Focused short term intervention (8-12 sessions)

SUMMARY:
The purpose of this study is to perform an evaluation of a trauma-focused short-term intervention (Narrative Exposure Therapy; Schauer, M., Neuner, F. & Elbert, T.) on a variety of clinical outcome measures (PTSD, Depression, Somatic Complaints, Dissociation) in women after sexual exploitation and women trafficking.

ELIGIBILITY:
Inclusion Criteria:

* Sexual Exploitation or Women Trafficked or Forced Prostitution
* Symptoms of Post Traumatic Stress Disorder

Exclusion Criteria:

* Current Psychotic Symptoms

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-06; Primary Completion 2010-01 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
PTSD, Depression, Somatic Complaints, Dissociation | Pre-Test, 4-weeks-Post-Test, 6-months-follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Research and Psychological Outpatient Clinic, University of Konstanz, Center for Psychiatry, House 22, Konstanz, Germany